CLINICAL TRIAL: NCT01212367
Title: A Pilot Study of Repeated Dose Intrapleural Adenoviral-Mediated Interferon-Alpha (SCH 721015, Ad.hIFN-a2b) Gene Transfer for Malignant Pleural Mesothelioma
Brief Title: Intrapleural Gene Transfer for Pleural Mesothelioma
Acronym: IFN-alpha
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 18508; 808806; P01CA066726 (NIH)
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: Gene transfer; Immunology; Cancer
MeSH Terms: conditions — Mesothelioma, Malignant; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dose Level 1 (Experimental)
  Interventions: Biological: SCH 721015
- Dose Level 2 (Experimental): This is a dose de escalation.
  Interventions: Biological: SCH 721015

INTERVENTIONS:
Biological: SCH 721015 — 1.0 x 10e12 viral particles on Days 1 and 4
  Other Names: Adenoviral-mediated Interferon-alpha; Ad.IFN-alpha
  Arms: Dose Level 1
Biological: SCH 721015 — 3.0 x 10e11 viral particles on Days 1 and 4
  Other Names: Adenoviral-mediated Interferon-alpha; Ad.IFN-alpha
  Arms: Dose Level 2

SUMMARY:
This research will study how to activate the immune system by using gene transfer. Gene transfer involves inserting a specially designed gene into cancer cells. A gene is a part of the genetic code that instructs the cells of our bodies to produce specific compounds (proteins) important for the makeup or function of the cell. The study hypothesis is that repeated doses of SCH 721015 given over a three day interval would result in gene transfer.

DETAILED DESCRIPTION:
Ad.hIFN-α (SCH 721015, adenoviral-mediated interferon alpha) is a replication-defective recombinant adenoviral vector containing the human interferon-alpha (hIFN-alpha) gene. This Phase I study is designed to evaluate the safety and maximum tolerated dose (MTD) of two doses of Ad.hIFN-alpha injected into the pleural (intrapleural, IP) and given 4 days apart in subjects with pleural mesothelioma.

Subjects who meet eligibility will have a pleural catheter placed 2 weeks prior to the first dose. Subjects are then admitted to the research center on Days 1 and 4 for dosing and overnight observation. Subjects are then followed-up as outpatients for a total of 6 months. Radiographic evaluations are repeated on Day 64 and at 6 months. The pleural catheter is removed once it is not necessary.

ELIGIBILITY:
Inclusion Criteria:

* evidence of progressive disease after standard first line treatment of mesothelioma; OR patient has refused standard first line treatment of mesothelioma
* evaluable disease
* No radiotherapy and/or treatment with chemotherapeutic, cytotoxic, or immunologic agents within 14 days prior to infusion of the IFN-α vector
* Must have a pleural space involved with tumor accessible for pleural catheter insertion
* FEV1> 1 liter or 40% of predicted value
* Must have an anti-adenoviral neutralizing antibody titer equal to or less than 1:1000. This will be measured by the Penn Vector Core

Exclusion Criteria:

* Presence of HIV or Hepatitis B infection
* Use of concurrent systemic steroids, immunosuppressives, or any other medications that can directly or indirectly suppress the immune system
* Presence of any other life-threatening illness, such as unstable angina, severe oxygen dependence, significant chronic obstructive pulmonary disease (COPD), end stage liver or renal disease
* Presence of untreated brain metastases
* Prior bone marrow or stem cell transplants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
To analyze gene transfer with two does separated by three-day interval | After the first dose and at each visit until day 94

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sterman, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Sterman DH, Haas A, Moon E, Recio A, Schwed D, Vachani A, Katz SI, Gillespie CT, Cheng G, Sun J, Papasavvas E, Montaner LJ, Heitjan DF, Litzky L, Friedberg J, Culligan M, June CH, Carroll RG, Albelda SM. A trial of intrapleural adenoviral-mediated Interferon-alpha2b gene transfer for malignant pleural mesothelioma. Am J Respir Crit Care Med. 2011 Dec 15;184(12):1395-9. doi: 10.1164/rccm.201103-0554CR. Epub 2011 Jun 3. PMID 21642245